CLINICAL TRIAL: NCT04472533
Title: Role of Inflammation and Angiogenesis in Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Serum Bio-markers in Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: T01502
Record Dates: First submitted 2020-07-06; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Hypertension, Primary, 4
Keywords: inflammation; angiogenesis
MeSH Terms: conditions — Hypertension, Pulmonary; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CTEPH: Patients diagnosed with chronic thromboembolic pulmonary hypertension
- CTED: Patients diagnosed with chronic thromboembolic disease but no evidence of pulmonary hypertension
- Control: Healthy control subjects

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is caused by scarred blood clots in the blood vessels supplying the lungs. This in turn leads to failure of the right side of the heart. The reason why these scarred clots form is unknown. An operation to remove the scarred clots, known as pulmonary endarterectomy, is a potential cure. However, some patients have persistent obstructions within the blood vessels and heart failure even after surgery.

It is thought that abnormal levels of proteins, found in the blood stream and responsible for inflammation and the development of new blood vessels may have role in causing the disease. In this study, these proteins were measured to assess whether they provide clues as to the cause of the disease and whether they could be used for the risk stratification of patients.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is an underdiagnosed form of pulmonary hypertension whose pathogenesis remains to be fully elucidated. Altered endothelial homeostasis, defective angiogenesis and inflammation have been implicated. The formation of the organised occlusions is considered to arise from a failure to resolve acute pulmonary emboli. There is emerging evidence supporting the role of mediators of angiogenesis, inflammation and the coagulation cascade (and their many interactions) in CTEPH. Pulmonary endarterectomy (PEA), to remove these occlusions, may be a cure in some patients. Assessing circulating proteins associated with these processes may be not only useful for understanding disease pathogenesis but may also lead to improvements in clinical assessment.

The study was approved by the Regional Ethics Committee (Papworth Hospital Research Tissue Bank; 08/H0304/56+5). Consecutive patients undergoing PEA surgery at Royal Papworth Hospital National Health Service Foundation Trust, United Kingdom, who consented for participation in the Research Tissue Bank between February 2012 and August 2014, were recruited. A validation data set included all consecutive samples collected from CTEPH patients prior to PEA between April 2010 and Aug 2017. Patients were diagnosed in accordance with international guidelines.

Patients had serum samples collected from a peripheral vein prior to PEA. In a subset of patients, further sampling was performed at the first follow up visit to Papworth Hospital 3-6 months post-PEA. Customized human cytokine/chemokine magnetic bead assays and customized human angiogenesis/growth factor assays were used to measure levels of circulating proteins in these serum samples (interleukin [IL] 6, IL8, IL10, tumour necrosis factor [TNF] α, angiopoietin 2 [Ang2], endoglin, vascular endothelial growth factor [VEGF] a, VEGFc, VEGFd and bone morphogenetic protein 9 [BMP9]).

Levels were compared to levels from patients with chronic thromboembolic disease but no pulmonary hypertension (CTED) and healthy age and sex matched controls. In addition multivariate rank regression models were used to assess associations between levels of circulating proteins and clinical assessments carried out as part of the patients routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give informed written consent
* Patients diagnosed with chronic thromboembolic pulmonary hypertension (CTEPH) according to international guidelines at an expert pulmonary hypertension centre
* Patients diagnosed with chronic thromboembolic disease (CTED) according to international guidelines at an expert pulmonary hypertension centre
* Age and sex matched healthy volunteers

Exclusion Criteria:

* Patients with inflammatory comorbidities
* Patients taking immunosuppressant medication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with CTEPH, CTED and healthy control volunteers at the Royal Papworth Hospital.
Sampling Method: Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Assess the differences between circulating biomarkers between patients with CTEPH, CTED and controls | 24 hours
  Assess differences in inflammatory cytokines (IL6, 8, 10, TNFa, hsCRP [all measured in pg/ml]) and markers of angiogenesis (Ang2, BMP9, Endoglin, VEGFa, VEGFc, VEGFd [all measured in pg/ml]) in patients with CTEPH compared to healthy controls

SECONDARY OUTCOMES:
Assess associations, using multivariate regression modelling, between IL6 and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum IL6 and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between IL8 and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum IL8 and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between IL10 and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum IL10 and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between TNFa and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum TNFa and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between Ang2 and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum Ang2 and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between BMP9 and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum BMP9 and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between Endoglin and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum Endoglin and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between VEGFa and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum VEGFa and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between VEGFc and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum VEGFc and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between VEGFd and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum VEGFd and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.
Assess associations, using multivariate regression modelling, between hsCRP and clinical assessments made prior to pulmonary endarterectomy in patients with CTEPH | 24 hours
  Using multivariate rank regression modelling, associations between serum hsCRP and clinical assessments (pulmonary haemodynamics, functional class, six-minute walk test distance) performed in patients with CTEPH prior to pulmonary endarterectomy will be assessed. Adjustments will be made to correct for multiple testing.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Pepke-Zaba, PhD FRCP, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113